CLINICAL TRIAL: NCT00644657
Title: The Effect of Clopidogrel on Coated-Platelets in Patients Undergoing Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13291
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Artery Disease; Chest Pain
Keywords: Platelets, platelet aggregation inhibitors
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clopidogrel — All subjects will receive a 300 mg loading dose
  Other Names: Plavix

SUMMARY:
This study will explore the effect of clopidogrel on coated-platelets in patients who are given a loading dose before diagnostic catheterization or percutaneous coronary intervention. We hypothesis that clopidogrel will reduce the percentage of platelets that are coated and therefore more hypercoagulable.

DETAILED DESCRIPTION:
Platelet activity will be determined by light transmission aggregometry at baseline, after a 300 mg dose of clopidogrel and after the catheterization and/or angioplasty procedure. The change in the percentage of platelets that are coated platelets will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients given clopidogrel loading dose before scheduled catheterization or percutaneous intervention

Exclusion Criteria:

* Acute coronary syndrome
* Unable to tolerate clopidogrel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliot Schechter, MD, Principal Investigator — University of Oklahoma
Locations (1):
- VA Medical Center, 1F187, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for cardiac catheterization and possible percutaneous intervention who received a loading dose of 300 mg of clopidogrel were recruited.
Groups:
- Clopidogrel Loading Dose: All subjects received a 300 mg loading dose of clopidogrel
Period: Overall Study
Arm/Group | Clopidogrel Loading Dose
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Clopidogrel: All 27 subjects received a 300 mg loading dose of clopidogrel
Arm/Group | Clopidogrel
Number analyzed (Participants) | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 25
The percentage of platelets that are "coated-Platelets" as measured by dual-agonist stimulation [Mean (Standard Deviation); unit: percent coated platelets] — In each patient the percentage of platelets that are collagen coated will be measured in each patient before clopidogrel administration.
  percent coated platelets | 40.0 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Coated Platelets After the Administration of Clopidogrel in Patients Undergoing Cardiac Catheterization and/or Angioplasty
Description: The percentage of platelets that are collagen coated after the administration of clopidogrel.
Time Frame: 24 hours after the administration of clopidotrel
Measure: Mean (Standard Deviation); unit: Percent of platelets that are coated.
Arm/Group | Clopidogrel Loading Dose
Number analyzed (Participants) | 27
Percent of platelets that are coated. | 32.8 (13.6) [0 to 0]

2. Secondary Outcome: The Percentage of Coated Platelets After Coronary Angiography and/or PCI
Description: The percentage of coated platelets 24 hours after coronary angiography and/or PCI
Time Frame: 6 hrs after procedure
Measure: Mean (Standard Deviation); unit: Percentage of platelets that are coated
Arm/Group | Clopidogrel Loading Dose
Number analyzed (Participants) | 27
Percentage of platelets that are coated | 33.9 (12.3)

ADVERSE EVENTS:
Arm/Group | Clopidogrel Loading Dose
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
Limited to primarily Male VA population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No